CLINICAL TRIAL: NCT04433910
Title: A Randomized, Prospective, Open Label Clinical Trial on the Use of Convalescent Plasma Compared to Best Supportive Care in Patients With Severe COVID-19
Brief Title: A Clinical Trial of Convalescent Plasma Compared to Best Supportive Care for Treatment of Patients With Severe COVID-19
Acronym: CAPSID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Deutsches Rotes Kreuz DRK-Blutspendedienst Baden-Wurttemberg-Hessen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAPSID2020-DRK-BSD; 2020-001310-38 (EudraCT Number)
Record Dates: First submitted 2020-05-06; First posted 2020-06-16 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma (Experimental): Convalescent plasma transfusion on day 1, 3 and 5.
  Interventions: Drug: Convalesscent Plasma
- Best supportive care (No Intervention): Best supportive care, cross over for patients with progressive disease on day 14 with convalescent plasma transfusion on day 15, 17 and 19.

INTERVENTIONS:
Drug: Convalesscent Plasma — Transfusion
  Arms: Convalescent plasma

SUMMARY:
This is a randomized, prospective, multicenter, open label clinical trial of convalescent plasma compared to best supportive care for treatment of patients with severe COVID-19.

The aim of the study is to explore the therapeutic effect of convalescent plasma transfusions on the survival and course of disease of patients with severe COVID-19. Convalescent plasma will be collected from recovered COVID-19 patients.

Patients with severe COVID-19 will be randomly assigned to two groups. Patients in the treatment group will receive covalescent plasma (250 - 325 ml) on days 1, 3 and 5. Patients in the control group will receive best supportive care. Clinical condition in all patients will be evaluated on day 14. In case of progressive COVID-19 on day 14 compared to baseline, patients in the control group may be switched to treatment with convalescent plasma on days 15, 17 and 19.

Fifty-three patients will be included in each group. Data of each patient will be collected until discharge but nor longer than day 60.

DETAILED DESCRIPTION:
This is a randomized, prospective, multicentre, open label clinical trial of convalescent plasma compared to best supportive care for treatment of patients with severe COVID-19.

The primary Endpoint is a dichotomous composite endpoint of survival and no longer fulfilling criteria of severe COVID-19 within 21 days after randomization. All criteria must be met in order to fulfil the primary endpoint.

Key secondary endpoints are time to clinical improvement (defined as time from randomization to an improvement of two points on the WHO R&D Blueprint seven-category ordinal scale for clinical improvement), the frequency and severity of adverse events and the case fatality rate on day 21, 35 and 60. Further secondary endpoints refer to the course of anti-SARS-CoV-2 antibodies in plasma donors and treated patients and the impact of donor criteria on the effectiveness of plasma units.

Patients with severe COVID-19 defined by a respiratory rate ≥ 30 breaths / minute under ambient air or the requirement of any type of ventilation support or the need for ICU treatment can be included in the trial. It is planned to enrol 106 patients. Patients will be stratified according to ventilation support and/or extracorporeal oxygenation and/or ICU treatment and will be equally asigned to two groups. The treatment group receives convalescent plasma (250 - 325 ml) on day 1, 3 and 5 and the control group will receive best supportive care. Clinical condition in all patients will be evaluated on day 14. In case of progressive COVID-19 on day 14 compared to baseline (i.e. day 0), patients in the control group may be switched to treatment with convalescent plasma on days 15, 17 and 19. A patient switching from the control group to convalescent plasma group because of progressive COVID-19 on day 14 will be considered as failure of the primary endpoint at final evaluation of the primary endpoint on day 21.

ELIGIBILITY:
Inclusion Criteria:

Patients with SARS-CoV-2 infection and

1. age ≥ 18 years and ≤ 75 years
2. SARS-CoV-2 infection confirmed by PCR (BAL, sputum, nasal and/or pharyngeal swap)
3. severe disease defined by at least one of the following:

   1. respiratory rate ≥ 30 breaths / minute under ambient air
   2. requirement of any type of ventilation support
   3. needs ICU treatment
4. Written informed consent by patient or legally authorized representative

Exclusion Criteria:

1. Accompanying diseases other than COVID-19 with an expected survival time of less than 12 months.
2. Previous treatment with any SARS-CoV-2-convalescent plasma
3. In the opinion of the clinical team, progression to death is imminent and inevitable within the next 48 hours, irrespective of the provision of treatment
4. Interval > 72 hours since start of ventilation support
5. Not considered eligible for extracorporeal oxygenation support (even in case of severe ARDS according to Berlin classification with Horovitz-Index < 100 mg Hg)
6. Chronic obstructive lung disease (COPD), stage 4
7. Lung fibrosis with UIP pattern in CT und severe emphysema
8. Chronic heart failure NYHA >= 3 and/or pre-existing reduction of left ventricular ejection fraction to ≤ 30%
9. Shock of any type requiring ≥ 0.5 µg/kg/min noradrenaline (or equivalent) or requiring more than two types of vasopressor medication for more than 8 hours
10. Liver cirrhosis Child C
11. Liver failure: Bilirubin > 5xULN and elevation of ALT /AST (at least one >10xULN).
12. Any history of adverse reactions to plasma proteins
13. Known deficiency of immunoglobulin A
14. Pregnancy
15. Breastfeeding women
16. Volume overload until sufficiently treated
17. Participation in another clinical trial with an investigational medicinal product

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of survival and no longer fulfilling criteria of severe COVID-19. | Day 21
  Dichotomous composite endpoint of survival and no longer fulfilling criteria of severe COVID-19. All criteria must be met in order to fulfil the primary endpoint.

SECONDARY OUTCOMES:
Time to clinical improvement | day 0 to discharge within a 60 day period
  Time to clinical improvement (defined as days from randomization to an improvement of two points on the WHO R&D Blueprint seven-category ordinal scale for clinical improvement) (Key secondary endpoint)
Frequency and severity of adverse events by CTCAE v5.0, (Key secondary endpoint) | day 0 to discharge within a 60 day period
Case fatality rate | on day 21, 35 and 60
Length of hospital stay Length of hospital stay (if applicable) | day 0 to 60
Length of stay in ICU | day 0 to 60
Duration of ventilation support / ECMO | day 0 to 60
Time until negative SARS-CoV-2 PCR (nasopharyngeal sample) | day 0 to 60
  time to first negative PCR will be assessed
Predictive value of comorbidities | day 0 to 60
  Comorbidities will be assessed and correlated to clinical improvement (WHO scale), mortality, length of stay in ICU (days) and length of hospital stay (days)
Predictive value of coagulation markers | day 0 to 60
  Correlation of coagulation markers (D-Dimers, prothrombin time, Partial Thromboplastin Time, ATIII, Fibrinogen) with clinical improvement (WHO scale), mortality, length of stay in ICU (days) and length of hospital stay (days)
Predictive value of inflamation | day 0 to 60
  Corelation of Inflammation (laboratory testing: CRP, IL-6, Ferritin, Blood cell Count) with clinical improvement (WHO scale), mortality, length of stay in ICU (days) and length of hospital stay (days)
Percentage of former COVID-19 patients willing to donate qualifying for plasma donation. | through study completion, an average of 8 months
Amount of Plasma Units that could be collected for the clinical trial | through study completion, an average of 8 months
Titer of anti-SARS-CoV-2 in transfused plasma units | any plasmaphereseis, through study completion, an average of 8 months
Impact of donor characteristics on anti-SARS-CoV-2 humoral response | up to 60 days
  Anti-SARS-CoV-2-antibody titers will be correlated with age; gender; severity of COVID-19; interval between resolution of symptoms and plasmapheresis of plasma donors
Course of anti-SARS-CoV-2 titer in both patient groups at different time points related to transfusion of convalescent plasma | up to 60 days
  Neutralizing anti-SARS-CoV-2 titers were measured by PRNT
Correlation of anti-SARS-CoV-2 titer in transfused plasma units and primary and key secondary outcomes. | day 0 to 60
  Correlation of antibody titers with: 1. "Survival and no longer fulfilling criteria of severe COVID-19"; 2. Change in WHO ordinal scale; 3. Time to clinical improvement; 4. Length of hospital stay; 5. Length of ICU stay; 6. Length of mechanical Ventilation or ECMO support.
Effect of timing of plasma transfusions | day 0 to 60
  Effect of timing of plasma transfusions on outcome: comparison of early treatment, i.e. day 1, 3 and 5 in convalescent plasma group vs. delayed treatment, i.e. day 15, 17, 19 in patients crossing over from control group due to progressive disease on day-14 assessment.
Long term survival | 15 month
  Long term survival up to 15 months after randomisation (patients in CCP group* compared to control group) or first plasma donation (CCP donors). And high-titer group versus low -titer group versus control.
Frequency of long COVID-19 | 15 month
  Frequency of long COVID-19* up to 15 months after randomisation (patients in CCP group* compared to control group) or first plasma donation (CCP donors).And high-titer group versus low -titer group versus control.
Resolution of pneumonia and functional recovery | 15 month
  Resolution of pneumonia and functional recovery* in patients (CCP group compared to control group and donors). Assessment will be done by CTCAE 5.0 and structured interview. And high-titer group versus low -titer group versus control.
Patient Reported Outcome: FACIT Fatigue Score | 15 month
  FACIT Fatigue Score: 0-53 : The higher the score, the better the quality of life Comparisons between patients CCP group compared to control group and donors and high-titer group versus low -titer group versus control group.
Patient Reported Outcome: FACIT Dyspnea Score | 15 month
  FACIT Dyspnea Score 1 and 2: 0-30 : The lhigher the score the worse is the dypnea Comparisons between patients CCP group compared to control group and donors and high-titer group versus low -titer group versus control group.
Patient Reported Outcome: EQ-5D-5L visual Scale | 15 month
  EQ-5D-5L visual scale: 0-100, The lower the socre, the worse is the health state Comparisons between patients CCP group compared to control group and donors and high-titer group versus low -titer group versus control group.
Patient Reported Outcome:EQ-5D-5L cross walk | 15 month
  EQ-5D-5L cross walk score: 0-1.0 The lower the socre, the worse is the health state Comparisons between patients CCP group compared to control group and donors and high-titer group versus low -titer group versus control group.
Laboratory markers: D-Dimers | 15 month
  D-Dimers will be correlated with the Levels of SARS-CoV-2 antodies as a measure of anti-SARS-CoV-2 immunity and compared between the patient groups (in patients: CCP group compared to control group and donors). The effect of SARS-CoV-2 vaccination* in control group, CCP group and CCP donors will also be taken into account.Measures will also be compeared between high-titer group versus low -titer group versus control group.
Laboratory markers: Fibrinogen | 15 month
  Fibronogen will be correlated with the Levels of SARS-CoV-2 antodies as a measure of anti-SARS-CoV-2 immunity and compared between the patient groups (in patients: CCP group compared to control group and donors). The effect of SARS-CoV-2 vaccination* in control group, CCP group and CCP donors will also be taken into account.Measures will also be compeared between high-titer group versus low -titer group versus control group.
Laboratory markers: CRP | 15 month
  CRP will be correlated with the Levels of SARS-CoV-2 antodies as a measure of anti-SARS-CoV-2 immunity and compared between the patient groups (in patients: CCP group compared to control group and donors). The effect of SARS-CoV-2 vaccination* in control group, CCP group and CCP donors will also be taken into account.Measures will also be compeared between high-titer group versus low -titer group versus control group.
Laboratory markers: Ferritin | 15 month
  Ferritin will be correlated with the Levels of SARS-CoV-2 antodies as a measure of anti-SARS-CoV-2 immunity and compared between the patient groups (in patients: CCP group compared to control group and donors). The effect of SARS-CoV-2 vaccination* in control group, CCP group and CCP donors will also be taken into account.Measures will also be compeared between high-titer group versus low -titer group versus control group.
Laboratory markers: IL-6 | 15 month
  IL-6 will be correlated with the Levels of SARS-CoV-2 antodies as a measure of anti-SARS-CoV-2 immunity and compared between the patient groups (in patients: CCP group compared to control group and donors). The effect of SARS-CoV-2 vaccination* in control group, CCP group and CCP donors will also be taken into account.Measures will also be compeared between high-titer group versus low -titer group versus control group.
Severity of long COVID-19 | 15 month
  Severity of long COVID-19* up to 15 months after randomisation (patients in CCP group* compared to control group) or first plasma donation (CCP donors). Grading according Post-COVID-19 Scale from 0 (no functional limitations) to 4 (severe functional limitations). Measures will also be compeared between high-titer group versus low -titer group versus control group.
Duration of long COVID-19 | 15 month
  Duration of long COVID-19* up to 15 months after randomisation (patients in CCP group* compared to control group) or first plasma donation (CCP donors). Measures will also be compeared between high-titer group versus low -titer group versus control group.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Schrezenmeier, Prof.Dr., Principal Investigator — IKT Ulm; Erhard Seifried, Prof.Dr.Dr., Study Director — German Red Cross Blood Service
Locations (16):
- Germany (16):
  - University Hospital Ulm, Ulm, Baden-Württmberg
  - University Hopsital Frankfurt, Frankfurt, Hessia
  - Saarland University Hospital, Homburg, Saarland
  - University Hospital Berlin, Charite, Berlin
  - Universitiy Hospital Dresden, Dresden
  - University Düsseldorf, Düsseldorf
  - University Hospital Freiburg, Freiburg im Breisgau
  - University Hospital Gießen, Giessen
  - University Hopsital Greifswald, Greifswald
  - Städtisches Klinikum Karslruhe, Karlsruhe
  - Universtity Hospital Schleswig-Holstein, Kiel
  - Universtity Hospital Schleswig-Holstein, Lübeck
  - University Hospital Mannheim, Mannheim
  - University Hospital Marburg, Marburg
  - Klinikum Stuttgart, Stuttgart
  - University Hospital Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Korper S, Gruner B, Zickler D, Wiesmann T, Wuchter P, Blasczyk R, Zacharowski K, Spieth P, Tonn T, Rosenberger P, Paul G, Pilch J, Schwable J, Bakchoul T, Thiele T, Knorlein J, Dollinger MM, Krebs J, Bentz M, Corman VM, Kilalic D, Schmidtke-Schrezenmeier G, Lepper PM, Ernst L, Wulf H, Ulrich A, Weiss M, Kruse JM, Burkhardt T, Muller R, Kluter H, Schmidt M, Jahrsdorfer B, Lotfi R, Rojewski M, Appl T, Mayer B, Schnecko P, Seifried E, Schrezenmeier H. One-year follow-up of the CAPSID randomized trial for high-dose convalescent plasma in severe COVID-19 patients. J Clin Invest. 2022 Dec 15;132(24):e163657. doi: 10.1172/JCI163657. PMID 36326824
- [Derived] Korper S, Schrezenmeier EV, Rincon-Arevalo H, Gruner B, Zickler D, Weiss M, Wiesmann T, Zacharowski K, Kalbhenn J, Bentz M, Dollinger MM, Paul G, Lepper PM, Ernst L, Wulf H, Zinn S, Appl T, Jahrsdorfer B, Rojewski M, Lotfi R, Dorner T, Jungwirth B, Seifried E, Furst D, Schrezenmeier H. Cytokine levels associated with favorable clinical outcome in the CAPSID randomized trial of convalescent plasma in patients with severe COVID-19. Front Immunol. 2022 Oct 6;13:1008438. doi: 10.3389/fimmu.2022.1008438. eCollection 2022. PMID 36275695
- [Derived] Korper S, Weiss M, Zickler D, Wiesmann T, Zacharowski K, Corman VM, Gruner B, Ernst L, Spieth P, Lepper PM, Bentz M, Zinn S, Paul G, Kalbhenn J, Dollinger MM, Rosenberger P, Kirschning T, Thiele T, Appl T, Mayer B, Schmidt M, Drosten C, Wulf H, Kruse JM, Jungwirth B, Seifried E, Schrezenmeier H; CAPSID Clinical Trial Group. Results of the CAPSID randomized trial for high-dose convalescent plasma in patients with severe COVID-19. J Clin Invest. 2021 Oct 15;131(20):e152264. doi: 10.1172/JCI152264. PMID 34464358
- [Derived] Conzelmann C, Gilg A, Gross R, Schutz D, Preising N, Standker L, Jahrsdorfer B, Schrezenmeier H, Sparrer KMJ, Stamminger T, Stenger S, Munch J, Muller JA. An enzyme-based immunodetection assay to quantify SARS-CoV-2 infection. Antiviral Res. 2020 Sep;181:104882. doi: 10.1016/j.antiviral.2020.104882. Epub 2020 Jul 29. PMID 32738255